CLINICAL TRIAL: NCT05958849
Title: A Single-arm, Open, Single-center Clinical Study of Sovalutinib in Combination With Solutumab and Tegeo in Second and Second Line for Advanced Pancreatic Cancer
Brief Title: Advanced Pancreatic Cancer
Acronym: PaC
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Zhejiang Cancer Hospital (Other)
Responsible Party: Principal Investigator, Luo Cong, Deputy Director, Zhejiang Cancer Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB-2023-277
Record Dates: First submitted 2023-06-08; First posted 2023-07-25 (Actual); Last update posted 2023-07-25 (Actual); Status verified 2023-07

CONDITIONS: Progression-free Survival

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Prospective Research (Experimental): Soventinib in combination with solutumab and tegeo dosing regimen:
  * Soventinib: 200 mg orally, within 1 hour of breakfast, administered once daily as a continuous dose, d1-d21, every 3 weeks in treatment cycles
  * Slulizumab: 300 mg administered intravenously, d1, every 3 weeks for one treatment cycle.
  * Tegeo: 40-60 mg/dose administered twice daily, d1-d14, continuously (dosing based on body surface area (BSA): 40 mg/dose for BSA ≤ 1.25 m2; 50 mg/dose for 1.25 ≤ BSA < 1.5 m2 and 60 mg/dose for BSA ≥ 1.5 m2), every 3 weeks for one treatment cycle. Dose adjustments, including suspension, dose reduction, or permanent discontinuation, were allowed as required by the protocol.
  Interventions: Drug: Sovalteinib Solutumab Tegeo

INTERVENTIONS:
Drug: Sovalteinib Solutumab Tegeo — Soventinib in combination with solutumab and tegeo for advanced pancreatic cancer

SUMMARY:
This study is a single-arm, open, single-center clinical study to observe and evaluate the efficacy and safety of sovalteinib in combination with solutumab and tegeo in second-line and post-line treatment of patients with advanced pancreatic cancer.

A total of 30 patients were enrolled in this study, which was divided into 3 phases: screening phase, treatment phase and follow-up phase. During the treatment period, tumor status was evaluated by imaging methods every 6 weeks (±7 days) until disease progression (PD, RECIST 1.1) or death (during patient treatment) or intolerable toxicity, and tumor treatment and survival status after disease progression were recorded. Safety observations included AE, changes in laboratory test values, vital signs, and changes in ECG. In addition, 10 ml of blood was drawn for testing in our laboratory before each treatment and at the time of disease progression before the patients were enrolled, and the exploration of the efficacy-related biomarker BRCA1 was performed by blood samples.

ELIGIBILITY:
Inclusion Criteria:

Subjects must meet all of the following conditions for enrollment:

1. subjects voluntarily enrolled in this study and signed an informed consent form, with good compliance and cooperation with follow-up;
2. patients with unresectable focally advanced or metastatic pancreatic cancer diagnosed by pathological histology or cytology
3. age between 18 and 75 years (both 18 and 75 years), male or female
4. ECOG score: 0-1; expected survival ≥ 12 weeks;
5. have progressed after receiving at least one prior systemic therapy for locally progressive or metastatic pancreatic cancer (including patients on first- or second-line regimens containing 5-FU)
6. have at least one measurable lesion (according to RECIST 1.1 criteria); ≥ 10 mm in diameter as accurately measured by magnetic resonance imaging (MRI) enhancement or computed tomography (CT) enhancement, and at least 20 mm in diameter as determined by conventional CT scan
7. no serious organic diseases of the heart, lungs, brain and other organs;
8. essentially normal function of major organs and bone marrow:

   1. routine blood (no blood transfusion, no granulocyte colony-stimulating factor [G-CSF], no drug correction within 14 days prior to screening): leukocytes ≥ 4.0 x 109/L, neutrophils ≥ 1.5 x 109/L, platelets ≥ 80 x 109/L, hemoglobin ≥ 90 g/L;
   2. International normalized ratio (INR) and activated partial thromboplastin time (APTT ) ≤ 1.5 x upper limit of normal (ULN);
   3. liver function (no albumin transfusion within 14 days prior to screening): serum total bilirubin ≤ 1.5 x ULN, ALT/AST ≤ 3 x ULN, and serum total bilirubin ≤ 1.5 x ULN after internal/external drainage for obstructive jaundice;
   4. Renal function: serum creatinine ≤ 1.5 x ULN, creatinine clearance (CCr) ≥ 50 mL/min;
   5. normal cardiac function, two-dimensional cardiac ultrasound detection of left ventricular ejection fraction (LVEF ) ≥ 50%; New York Heart Association (NYHA) classification <3.
9. Male or female patients of childbearing potential voluntarily use an effective contraceptive method such as a double barrier method, condom, oral or injectable contraceptive medication, IUD, etc. during the study period and within 6 months of the last study dose. All female patients will be considered fertile unless the female patient is spontaneously menopausal, has undergone artificial menopause, or has been sterilized.

Exclusion Criteria:

1. participation in other antitumor drug clinical trials within 4 weeks prior to enrollment, including: interventional, chemotherapy, bioimmunotherapy, targeted therapy, etc;
2. previous treatment with a previous vascular endothelial growth factor (VEGFR) inhibitor or previous treatment with an immune checkpoint inhibitor, and previous treatment with tegeo;
3. other malignancies within the past 5 years, except for basal or squamous cell carcinoma of the skin after radical surgery, or carcinoma in situ of the cervix
4. patients who have developed any brain metastases or are currently developing brain metastases
5. with liver metastases representing 50% or more of the total liver volume as determined by the investigator
6. have undergone any surgery (other than biopsy) or invasive treatment or operation within 4 weeks prior to enrollment and the surgical incision has not fully healed (except for intravenous placement, puncture drainage, internal/external drainage procedures for obstructive jaundice, etc.)
7. have received local antitumor therapy such as hepatic artery interventional embolization, cryoablation of liver metastases or radiofrequency ablation within 4 weeks prior to enrollment;
8. clinically significant electrolyte abnormalities in the judgment of the investigator;
9. the patient has current hypertension that is not controlled by medication, specified as: systolic blood pressure ≥ 140 mmHg and/or diastolic blood pressure ≥ 90 mmHg
10. urine routine suggestive of urine protein ≥ 2+ and 24-hour urine protein amount > 1.0 g
11. patients whose tumors are judged by the investigator to be at high risk of invading important blood vessels and causing fatal hemorrhage during the follow-up study;
12. patients with evidence or history of significant bleeding tendency within 3 months prior to enrollment (bleeding >30 mL within 3 months with vomiting, black feces, blood in stool), hemoptysis (>5 mL of fresh blood within 4 weeks); those with a history of hereditary or acquired bleeding disorders or coagulation disorders, who have had clinically significant bleeding symptoms within 3 months or have a clear bleeding tendency, such as gastrointestinal bleeding, hemorrhagic gastric ulcers, etc;
13. clinically significant cardiovascular disease, including but not limited to acute myocardial infarction, severe/unstable angina, or coronary artery bypass grafting within 6 months prior to enrollment; congestive heart failure New York Heart Association (NYHA) class >2; ventricular arrhythmias requiring pharmacologic treatment; and electrocardiogram (ECG) showing QT c interval ≥480 ms;
14. active or uncontrolled serious infection (≥ CTCAE grade 2 infection);
15. unremitting toxic reactions above CTCAE grade 2 due to any prior anticancer therapy, excluding alopecia, lymphopenia and neurotoxicity ≤ grade 2 due to oxaliplatin;
16. women who are pregnant (positive pregnancy test prior to dosing) or breastfeeding
17. any other disease with a clinically significant metabolic abnormality, physical examination abnormality or laboratory test abnormality that, in the judgment of the investigator, gives reason to suspect that the patient has a disease or condition that is inappropriate for the use of the study drug (e.g., has seizures and requires treatment) or that would affect the interpretation of the study results or place the patient at high risk
18. known human immunodeficiency virus (HIV) infection; known history of clinically significant liver disease, including viral hepatitis [known hepatitis B virus (HBV) carriers must be excluded from active HBV infection, i.e., positive HBV DNA (>1×104 copies/mL or >2000 IU/ml); known hepatitis C virus infection (HCV) with HCV RNA positive (>1×103 copies/mL), or other hepatitis, cirrhosis];
19. persons with any active, known or suspected autoimmune disease (including but not limited to: myasthenia gravis, myositis, autoimmune hepatitis, systemic lupus erythematosus, rheumatoid arthritis, enterocolitis, multiple sclerosis, vasculitis, glomerulonephritis, uveitis, pituitary inflammation, hyperthyroidism, etc.)
20. those who are allergic or suspected to be allergic to the study drug or similar drugs
21. Patients who, in the judgment of the investigator, have other factors that could affect the outcome of the study or force the termination of this study midway, such as alcoholism, drug abuse, other serious illnesses (including psychiatric illnesses) requiring comorbid treatment, serious laboratory test abnormalities, accompanied by family or social factors that would affect the safety of the patient.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-08-01 (Estimated); Primary Completion 2024-07-01 (Estimated); Study Completion 2025-07-30 (Estimated)

PRIMARY OUTCOMES:
PFS | through disease progression, an average of 6 months
  Time between the start of treatment and the onset of (any aspect of) progression of the tumor or death (from any cause)

SECONDARY OUTCOMES:
ORR | through disease progression, an average of 6 months
  The proportion of patients whose tumor volume shrinks to a pre-specified value and who can maintain the minimum time requirement is the sum of the proportion in complete and partial remission.
DCR | through disease progression, an average of 6 months
  The number of cases that achieved remission (PR+CR) and stable lesions (SD) after treatment as a percentage of the evaluable cases.
OS | through patients' death, an average of 12 months
  Time from start of treatment to death (from any cause)

IPD SHARING:
Plan to Share IPD: No